CLINICAL TRIAL: NCT05707468
Title: Safety and Efficacy Study of Neoadjuvant Radiohormonal Therapy for Oligometastatic Prostate Cancer: a Multi-center Randomized Controlled Clinical Trial
Brief Title: Neoadjuvant Radiohormonal Therapy for Oligometastatic Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Director, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Changhai Hospital PCa
Record Dates: First submitted 2022-12-15; First posted 2023-02-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Oligometastatic Prostate Carcinoma
MeSH Terms: interventions — abiraterone

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio between arm A (hormone) and arm B (neoadjuvant hormone and RT).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (hormone) (Active Comparator): The patients in arm A with oligometastatic PCa will receive long-term ADT combined with abiraterone.
  Interventions: Drug: ADT combined with abiraterone
- B (neoadjuvant hormone and RT) (Experimental): The patients in arm B with oligometastatic PCa will receive 1 month of naADT, followed by metastasis-directed radiation and abdominal or pelvic radiotherapy. Then, radical prostatectomy will be performed at intervals of 5-15 weeks after radiotherapy, and long-term ADT will be continued.
  Interventions: Radiation: neoadjuvant hormone and RT

INTERVENTIONS:
Drug: ADT combined with abiraterone — The patients will receive long-term ADT combined with abiraterone.
  Arms: A (hormone)
Radiation: neoadjuvant hormone and RT — The patients will receive 1 month of naADT, followed by metastasis-directed radiation and abdominal or pelvic radiotherapy. Then, radical prostatectomy will be performed at intervals of 5-15 weeks after radiotherapy, and long-term ADT will be continued.
  Arms: B (neoadjuvant hormone and RT)

SUMMARY:
The optimal treatment for oligometastatic prostate cancer (OMPC) is still on its way. Accumulating evidence has proven the safety and feasibility of radical prostatectomy and local or metastasis-directed radiotherapy for oligometastatic patients. The aim of this trial is to compare the safety and feasibility outcomes of metastasis-directed neoadjuvant radiotherapy (naRT) and neoadjuvant androgen deprivation therapy (naADT) followed by robotic-assisted radical prostatectomy (RARP) to ADT combined with abiraterone for treating OMPC.

DETAILED DESCRIPTION:
The present study will be conducted as a prospective, open-label, two arms clinical trial. Patients with ≤ 3 de novo oligometastatic PCa, diagnosed on Ga-68 prostate-specific membrane antigen (PSMA) PET/CT, will be randomized in a 1:1 ratio between arm A (hormone) and arm B (neoadjuvant hormone and RT). The patients in arm A with oligometastatic PCa will receive long-term ADT combined with abiraterone. The patients in arm B with oligometastatic PCa will receive 1 month of naADT, followed by metastasis-directed radiation and abdominal or pelvic radiotherapy. Then, radical prostatectomy will be performed at intervals of 5-15 weeks after radiotherapy, and long-term ADT will be continued. The primary endpoints of the study are progression-free survival (PFS) including biochemical recurrence-free survival (bPFS), and radiological progression-free survival (RPFS). The secondary endpoints include quality of life (QoL), time to CRPC, positive surgical margin (pSM), overall survival (OS), postoperative continence, and toxicities parameters.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate without small cell features
* Oligometastatic PCa assessed by Ga-68 prostate-specific membrane antigen (PSMA), PET/CT
* <4 bone oligometastases, lymph node metastasis below the renal artery level
* Expected survival time >5 years
* World Health Organization (WHO) performance status 0-1
* Be willing to give written informed consent.

Exclusion Criteria:

* Any previous or ongoing treatment for PCa, including radiotherapy, ADT, chemotherapy, focal treatment, etc.
* Patients who have previously undergone transurethral resection or enucleation of the prostate.
* Patients who have undergone other abdominal surgery within the last 3 months
* Patients who have visceral metastases
* Patients with a history of long-term anticoagulant use and anti-platelet drug use and who stopped anticoagulant therapy less than 1 week before registration
* Patients with other malignancies and acute or chronic infections such as human immunodeficiency virus (HIV) (+), hepatitis C virus (HCV) (+) and/or positive syphilis
* Severe or active comorbidities likely to impact the advisability of radiotherapy
* Any other serious underlying medical, psychiatric, psychological, familial, or geographical condition, which, according to the judgement of the investigator, may affect the planned staging, treatment and follow-up or patient compliance or may cause high-risk treatmentrelated complications for the patient
* Patients who have participated in other clinical trials within the last 3 months
* Patients who refuse to undergo RALP
* Patients unsuitable for participation in this clinical trial as per the judgement of the investigator.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival (PFS) | Assessment progression-free survival (PFS) at 3 years
  To assess progression-free survival (PFS) including biochemical recurrence-free survival (bPFS), and radiological progression-free survival (RPFS).

SECONDARY OUTCOMES:
quality of life (QoL) | through study completion, an average of 3 years
  quality of life (QoL)
time to castration-resistant prostate cancer (CRPC) | through study completion, an average of 3 years
  To assess the time to castration-resistant prostate cancer (CRPC)
5-year overall survival (OS) | Assessment overall survival (OS) at 5 years
  To assess the overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - First Affiliated Hospital and Medical College of Soochow University, Suzhou, Jiangsu
  - Jiangnan University Medical Center, Wuxi, Jiangsu
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - The Second Affiliated Hospital of Naval Medical University, Shanghai
  - The First Affiliated Hospital of Naval Medical University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data including baseline characteristics,treatment information and follow-up data on toxicity, survival and disease control will be shared.
Supporting Information: Study Protocol
Time Frame: Within 5 years after the publication of the study.
Access Criteria: Data may be shared with radiation oncologists and specialists in surgerywho are interested in examining the efficacy and toxicity of oligometastatic prostate cancer treated withneoadjuvant radiohormonal therapy or androgen deprivation therapy (ADT) combined with abiraterone. Detailed study protocol should be emailed along with the request of the data. We may carefully review the study protocol, and data will only be shared with well-designed studies.

REFERENCES:
- [Derived] Fan Z, Li D, Yan S, Zhao X, Yin L, Xu W, Wang Y, Zhang H, Chang Y, Ren S. NEoAdjuvant radiohormonal therapy versus standard of care for oligometastatic prostate cancer (NEAR-TOP): study protocol of a multicenter, open-label, randomised controlled trial. BMC Cancer. 2025 Apr 24;25(1):768. doi: 10.1186/s12885-024-13201-w. PMID 40275195